CLINICAL TRIAL: NCT07134621
Title: Target Organ Damage in Patients With Repaired Coarctation of Aorta and Exercise Induced Hypertension
Status: Enrolling by invitation | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Other Study IDs: 0120-135/2023/6
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Coarctation of the Aorta
MeSH Terms: conditions — Aortic Coarctation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to obtain data on the effect of exercise induced hypertension on target organs in adult patients with repaired coarctation of the aorta. The main questions it aims to answer are:

* patients with exercise induced hypertension have signs of hypertensive heart disease?
* patients with exercise induced hypertension have increased arterial stiffness?
* patients with exercise induced hypertension have signs of hypertensive renal damage? Participants will be invited for an outpatient appointment during which medical history and physical investigation will be performed. They will undergo cardiopulmonary exercise testing during which blood pressure will be measured regularly. Transthoracic echocardiography will also be performed as well as assessment of arterial stiffness by measuring pulse wave velocity. Renal function will be assessed by blood and urine analysis.

ELIGIBILITY:
Inclusion Criteria:

* adult patients aged 18 years and older
* history of coarctation of aorta repair

Exclusion Criteria:

* haemodynamically significant recoarctation
* arterial hypertension at rest
* antihypertensive therapy
* associated haemodynamically significant valvular heart disease
* associated complex congenital heart disease
* advanced heart failure
* symptomatic arrhythmias
* cognitive or physical limitations to perform exercise stress testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 years and older with repaired coarctation of aorta.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of patients with EIH who also have signs of hypertensive heart disease. | At enrolment.
Number of patients with EIH and increased arterial stiffness. | At enrolment.
Number of patients with EIH and signs of hypertensive renal damage. | At enrolment.

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Ljubljana, Ljubljana, Slovenia